CLINICAL TRIAL: NCT00340327
Title: An Ascending Single Dose Study of the Safety and Pharmacokinetics of IMA-638 Administered to Healthy Japanese Subjects
Brief Title: Study Evaluating IMA-638 in Healthy Japanese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3174K1-101
Record Dates: First submitted 2006-06-16; First posted 2006-06-21 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
Keywords: healthy subjects
MeSH Terms: interventions — anrukinzumab

INTERVENTIONS:
Drug: IMA-638

SUMMARY:
The purpose of this study is to evaluate the safety and drug levels for single, ascending doses of IMA-638 in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* First generation healthy Japanese men and women of non-childbearing potential.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-06; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety will be measured by evaluating physical examinations, vital signs, electrocardiograms (ECGs), and clinical laboratory test results.

SECONDARY OUTCOMES:
Drug levels and associated biomarkers will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Glendale, California, United States